CLINICAL TRIAL: NCT01113723
Title: A Randomized Prospective Study to Compare Tracheal Intubation With the CMAC Device to Fiberoptic Bronchoscopy in Patients With an Unstable Cervical Spine
Brief Title: Intubation of Patients With an Unstable Cervical Spine Using the CMAC Device
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Roya Yumul, M.D.,PhD., Residency program director, Department of anesthesiology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Pro00019845
Record Dates: First submitted 2010-04-23; First posted 2010-04-30 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-02

CONDITIONS: Laminectomy
Keywords: C-MAC; Fiberoptic bronchoscope; Laryngoscopy; Cervical spine injury; Glottic view; Tracheal intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CMAC Device (Other): CMAC Intubating device time to achieve successful tracheal intubation.
  Interventions: Device: CMAC
- Fiberoptic bronchoscope (Active Comparator): Fiberoptic bronchoscope Intubating device time to achieve successful tracheal intubation.
  Interventions: Device: Fiberoptic bronchoscope

INTERVENTIONS:
Device: Fiberoptic bronchoscope — Fiberoptic bronchoscope device
  Arms: Fiberoptic bronchoscope
Device: CMAC — CMAC Device
  Arms: CMAC Device

SUMMARY:
The purpose of this study is to evaluate whether tracheal intubation with the CMAC device decreases the time required for intubation as compared to intubation with the fiberoptic bronchoscope in patients with an unstable cervical spine. Both the CMAC device and the fiberoptic bronchoscope are currently commonly used in standard of care practices in the intubation of patients with cervical spine injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an unstable Cervical-spine as a result of C-spine injury.
* Patients scheduled to undergo inpatient surgical procedures under general anesthesia.
* Willingness and ability to sign an informed consent document.
* 18-80 years of age.
* ASA Class I - III adults of either sex

Exclusion Criteria:

* Patients deemed to be at significant airway risk to necessitate awake fiber optic intubation.
* Patients with a history of oral-pharyngeal cancer or reconstructive surgery.
* Emergency surgeries.
* Any other conditions which may interfere with the conduct of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roya Yumul, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CMAC Device: CMAC
  CMAC: CMAC Device
- Fiberoptic Bronchoscope: Fiberoptic bronchoscope device: the flexible fiberoptic scope (FFS)
Period: Overall Study
Arm/Group | CMAC Device | Fiberoptic Bronchoscope
Started | 70 | 70
Completed | 70 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fiberoptic Bronchoscope: Fiberoptic bronchoscope
  Fiberoptic bronchoscope: Fiberoptic bronchoscope device
- Total: Total of all reporting groups
Arm/Group | CMAC Device | Fiberoptic Bronchoscope | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (12) | 50 (12) | 53 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 38 | 70
  Male | 38 | 32 | 70
Region of Enrollment [Number; unit: participants]
  United States | 70 | 70 | 140

OUTCOME MEASURES:

1. Secondary Outcome: Time to Obtain Glottis Visualization (Seconds)
Description: Time to Obtain Glottis Visualization (Seconds): View of the glottis during the beginning of the intubation procedure. (approximately 1 minute) Glottic (the opening between the vocal cords at the upper part of the larynx) visualization comparison between the two devices in patients with an unstable cervical spine.
Time Frame: 1 minute
Population: Time to Obtain Glottis Visualization (Seconds) Glottic visualization during the beginning of the intubation procedure.
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Flexible Fiberoptic Scope (FFS): the flexible fiberoptic scope (FFS) : the flexible fiberoptic scope (FFS)
Arm/Group | CMAC Device | Flexible Fiberoptic Scope (FFS)
Number analyzed (Participants) | 70 | 70
Seconds | 32 (32) | 16 (14)

2. Primary Outcome: Intubation Time (Seconds)
Description: Times (seconds) following initial insertion of laryngoscope blade to placement of tracheal tube
Time Frame: 3 minutes
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | CMAC Device | Fiberoptic Bronchoscope
Number analyzed (Participants) | 70 | 70
Seconds | 35 (22) | 59 (36)

3. Primary Outcome: Time to Confirm the Placement of the Tracheal Tube
Description: It is the time (in seconds) following initial insertion of laryngoscope blade to confirm with CO2 waveform
Time Frame: up tp 3 minutes
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | CMAC Device | Fiberoptic Bronchoscope
Number analyzed (Participants) | 70 | 70
Seconds | 62 (31) | 99 (38)

ADVERSE EVENTS:
Groups:
- Flexible Fiberoptic Scope (FFS): the flexible fiberoptic scope (FFS) the flexible fiberoptic scope (FFS) : the flexible fiberoptic scope (FFS)
Arm/Group | CMAC Device | Flexible Fiberoptic Scope (FFS)
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No